CLINICAL TRIAL: NCT07170098
Title: Post-operative Pain Following Different Irrigation Activation and Disinfection Approaches in Single-rooted Teeth With Asymptomatic Apical Periodontitis: A Randomized Clinical Trial
Brief Title: Post-operative Pain After Different Irrigation and Disinfection Methods in Single-rooted Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Sema Sönmez Kaplan, Associate Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BİRUNİ-BAP-01-2023-01-05; BİRUNİ-BAP-01-2023-01-05 (Other Grant/Funding Number: Biruni University)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Pain; Apical Periodontitis; Asymptomatic Infections
Keywords: Asymptomatic apical periodontitis; Diode laser; EDDY; EndoActivator; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative; Periapical Periodontitis; Asymptomatic Infections | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: Parallel-group randomized controlled trial
Who Masked: Participant
Masking Description: Patients were blinded to the irrigation and disinfection method. The operator was not blinded due to the nature of the interventions. Post-operative pain was self-reported by patients using numerical rating scales and outcomes assesor was was not blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EDDY sonic irrigation (Experimental): Final irrigation activation was performed using the EDDY sonic system with 5.25% NaOCl for three 20-second cycles, followed by 17% EDTA for 30 seconds and 5 mL saline. No laser irradiation was applied.
  Interventions: Device: EDDY sonic irrigation system
- EndoActivator (EA) sonic irrigation (Experimental): Final irrigation activation was performed using the EndoActivator (EA) medium tip with 5.25% NaOCl for three 20-second cycles, followed by 17% EDTA for 30 seconds and 5 mL saline. No laser irradiation was applied.
  Interventions: Device: EndoActivator (EA) sonic irrigation system
- EDDY sonic irrigation + 980-nm diode laser (Experimental): Final irrigation activation was performed using the EDDY sonic system as in Arm 1, followed by adjunctive 980-nm diode laser irradiation (1.2 W, 50 Hz, 12 J per cycle, 4 cycles, pulsed mode).
  Interventions: Device: EDDY sonic irrigation system; Device: 980-nm diode laser
- EndoActivator (EA) sonic irrigation + 980-nm diode laser (Experimental): Final irrigation activation was performed using the EndoActivator (EA) system as in Arm 2, followed by adjunctive 980-nm diode laser irradiation (1.2 W, 50 Hz, 12 J per cycle, 4 cycles, pulsed mode).
  Interventions: Device: EndoActivator (EA) sonic irrigation system; Device: 980-nm diode laser

INTERVENTIONS:
Device: EDDY sonic irrigation system — Sonic activation of irrigating solutions during endodontic treatment.
  Arms: EDDY sonic irrigation; EDDY sonic irrigation + 980-nm diode laser
Device: EndoActivator (EA) sonic irrigation system — Sonic activation of irrigating solutions during endodontic treatment.
  Arms: EndoActivator (EA) sonic irrigation; EndoActivator (EA) sonic irrigation + 980-nm diode laser
Device: 980-nm diode laser — Diode laser irradiation during endodontic treatment.
  Arms: EDDY sonic irrigation + 980-nm diode laser; EndoActivator (EA) sonic irrigation + 980-nm diode laser

SUMMARY:
This randomized clinical trial aimed to evaluate post-operative pain (PP) in single-rooted teeth with asymptomatic apical periodontitis following final irrigation with sonic activation systems (EDDY and EndoActivator), with and without adjunctive 980-nm diode laser disinfection. Eighty patients were randomized into four groups: Group 1 (EDDY), Group 2 (EndoActivator), Group 3 (EDDY + laser), and Group 4 (EndoActivator + laser). PP intensity and analgesic intake were recorded at 8, 24, 48 hours, and on day 7. The study found no significant differences in PP or analgesic use among the groups, indicating that laser-assisted or different sonic activation methods did not reduce post-operative pain.

DETAILED DESCRIPTION:
Post-operative pain (PP) is a common concern following root canal treatment, influenced by mechanical, chemical, and microbial factors. Effective irrigation and disinfection are crucial to remove debris and microorganisms from complex canal systems. This study investigated the effects of two sonic irrigation activation systems, EDDY and EndoActivator (EA), with and without 980-nm diode laser disinfection, on PP in patients with single-rooted teeth diagnosed with asymptomatic apical periodontitis.

Eighty medically healthy adult patients (18-65 years) were randomly assigned to four groups. Group 1 underwent final irrigation with EDDY; Group 2 with EA; Group 3 with EDDY followed by laser irradiation; Group 4 with EA followed by laser irradiation. All procedures were completed in a single visit. PP was measured using a 0-10 numerical rating scale at 8, 24, 48 hours, and day 7. Analgesic consumption was also recorded.

Statistical analysis showed no significant differences among groups for age, sex, PP scores, or analgesic intake. None of the patients experienced severe pain or swelling requiring emergency intervention. The findings suggest that both EDDY and EA sonic irrigation systems, with or without adjunctive 980-nm diode laser disinfection, do not significantly affect post-operative pain or analgesic use following single-visit root canal treatment of asymptomatic apical periodontitis.

These results provide insight into the effectiveness of sonic irrigation activation and laser disinfection in routine endodontic practice, indicating that alternative techniques may be explored to optimize patient comfort and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy adult patients aged 18-65 years
* Patients diagnosed with asymptomatic apical periodontitis in permanent single-rooted teeth with closed apices and radiographic PAI score of 3 or 4
* Healthy periodontal conditions

Exclusion Criteria:

* Pregnant women
* Patients with systemic disorders
* Teeth with open apex, prosthetic restorations, mobility > grade I, periodontal pocket depth > 4 mm, non-restorable condition, calcified root canals, resorption, traumatic occlusion, or history of previous endodontic treatment
* Patients who had taken analgesics within 12 hours prior to intervention
* Patients who had received antibiotic therapy within the past month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Post-operative pain intensity | 8, 24, and 48 hours, and 7 days after the endodontic procedure
  Pain intensity was self-reported by patients using a numerical rating scale (0-10), where 0 indicates no pain and 10 indicates the worst possible pain.

SECONDARY OUTCOMES:
Analgesic consumption | 8, 24, and 48 hours, and 7 days after the endodontic procedure
  Patients recorded the type, dosage, and timing of analgesics taken during the postoperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No